CLINICAL TRIAL: NCT06298916
Title: A Phase 1/2a Study Utilizing 64Cu-LNTH-1363S (64Cu Radiolabeled FAPi PET/CT Imaging Agent) in Patients With Sarcoma or Gastrointestinal Tract Cancer (PHANTOM Trial)
Brief Title: 64Cu-LNTH-1363S in Patients With Sarcoma or Gastrointestinal Tract Cancer
Acronym: PHANTOM
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Lantheus Medical Imaging (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: FAPi-1301
Record Dates: First submitted 2024-02-22; First posted 2024-03-07 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-07

CONDITIONS: Metastatic Sarcoma; Esophageal Cancer; Gastric Cancer; Pancreatic Cancer; Colorectal Cancer; Sarcoma
Keywords: FAPi; Imaging; 64Cu-LNTH-1363S
MeSH Terms: conditions — Sarcoma; Esophageal Neoplasms; Stomach Neoplasms; Pancreatic Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Part 1: Metastatic Sarcoma Part 2: Non-metastatic sarcoma or gastrointestinal tract (GIT) cancer (esophageal, gastric, pancreatic, colorectal cancer)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Part 1 (Experimental): 6 patients will receive 8 ± 1 mCi (~90 μg mass dose) of the 64Cu-LNTH-1363S on Day 1 in the Intervention Period (raw data of each patient PET scan will be re-processed using a computer program to simulate scans of the same patient with 6 mCi and 4 mCi 64Cu injected activities).
  Interventions: Combination Product: 64Cu-LNTH-1363S
- Experimental Part 2 (Experimental): First 6 evaluable patients will receive the optimal radioactivity determined in Part 1. The remaining 14 evaluable patients will receive either the optimal radioactivity determined in Part 1 (if the sum of the average image quality scores of the first 6 patients is higher or equal to 10.5), or 8 ± 1 mCi (if the sum of the average image quality scores of the first 6 patients is less than 10.5).
  Interventions: Combination Product: 64Cu-LNTH-1363S

INTERVENTIONS:
Combination Product: 64Cu-LNTH-1363S — 64Cu-LNTH-1363S, is a highly selective, high affinity FAP inhibitor (FAPi) that is radiolabeled with Copper-64 (64Cu) for PET/CT Imaging,

SUMMARY:
This is a multicenter, open-label, prospective Phase 1/2a study to assess safety and tolerability, establish dosimetry and to identify an optimal imaging dose (radioactivity) and imaging time window of 64Cu-LNTH-1363S, and to compare its imaging biodistribution with FAP expression by IHC in patients with sarcomas or GIT cancers. The study will be conducted in 2 parts (Part 1 and Part 2).

DETAILED DESCRIPTION:
Part 1 will determine the biodistribution, dosimetry, optimal dose (radioactivity) and imaging time window of 64Cu-LNTH-1363S in 6 evaluable patients with supposed FAP-expressing solid tumors (metastatic sarcomas). All six patients will receive 8 ± 1 mCi (~90 μg mass dose) in this study. All images will undergo analysis by blinded central readers. Optimal radioactivity and timing window will be determined based on image quality scores and measured tumor-to-background ratio. Part 1 of the study will last approximately 3 weeks for each patient and includes a Screening Period (up to 14 days), a 1-day Intervention Period and a Safety Follow-up Period (7 days post dose).

Part 2 will evaluate 64Cu-LNTH-1363S correlation with FAP expression measured by IHC (SUVmax and SUVmean vs IHC score) in 20 evaluable patients with non-metastatic, operable, supposed FAP-expressing solid tumors (sarcomas, esophageal, gastric, pancreatic, colorectal) planned for surgery within 60 days (from study imaging). If the optimal radioactivity determined from Part 1 is less than 8 ± 1 mCi, the first 6 patients in Part 2 will be used to validate this optimal radioactivity.

Part 2 of the study will last approximately 10 to 11 weeks and includes: a Screening Period (up to 14 days), a 1-day Intervention Period, a 1 day Safety Followup Period (Day 2) and a Scheduled Surgery IHC Sample Collection Period (from Day 2 to Day 60).

Both Part 1 and Part 2 of the study will also monitor cardiac safety by detecting changes in HR, T wave, ST segment and other ECG parameters and characterizing the concentration-response relationship of 64Cu-LNTH-1363S for QT and corrected QT interval (QTc) prolongation.

ELIGIBILITY:
Inclusion Criteria: Part 1

Patients are eligible to be included in the study only if all of the following criteria apply:

1. Patient must be ≥ 15 years of age and must have provided written informed consent and assent, where applicable (by patient or legal guardian). Those aged ≥15 to <18 years must weigh at least 55 kg.
2. Patients with suspected FAP-expressing metastatic sarcoma.
3. Patients must have histological, pathological, and/or cytological confirmation of a metastatic sarcoma (e.g., undifferentiated pleomorphic sarcoma, liposarcoma, Leiomyosarcoma, myxofibrosarcoma, solitary fibrous tumor, Ewing's sarcoma, synovial sarcoma, sarcoma not otherwise specified, osteosarcoma).
4. Patients must be willing to consent to provide sufficient and adequate archived tumor tissue samples (formalin fixed, paraffin embedded sample), preferably from a biopsy of a tumor lesion obtained either at the time of or after the diagnosis of disease; if archival tissue sample is unavailable, a new biopsy should be performed on the most accessible lesion(s) to obtain the tumor tissue sample.
5. Adequate renal function as determined by a calculated creatinine clearance ≥ 60 mL/min (Cockcroft Gault equation).
6. Women of childbearing potential (WOCBP) must have a negative beta-human chorionic gonadotropin (β-hCG) test and must not be breastfeeding. WOCBP must agree to use a highly effective method of contraception during the study and for 28 days after the last injection of the study drug.
7. Male subjects who are able to father a child must agree to avoid impregnating a partner, to adhere to a highly effective method of contraception and to not donate sperm during the study and for 28 days after the last injection of the study drug.

Inclusion Criteria: Part 2

1. Patient must be ≥ 15 years of age and must have provided written informed consent and assent, where applicable (by patient or legal guardian). Those aged ≥15 to <18 years must weigh at least 55 kg.
2. Patients must have histological, pathological, and/or cytological confirmation of a sarcoma or GIT cancers e.g., esophageal, gastric, pancreatic, colorectal cancer.
3. Patients must have suspected FAP expressing sarcoma or GIT cancers and planned for surgery within 60 days (from study imaging).
4. Patients must be willing to consent to provide sufficient and adequate tumor tissue samples (formalin fixed, paraffin embedded sample), from their planned surgery after participating in study imaging.
5. Adequate renal function as determined by a calculated creatinine clearance ≥ 60 mL/min (Cockcroft Gault equation).
6. Women of childbearing potential (WOCBP) must have a negative beta-human chorionic gonadotropin (β-hCG) test and must not be breastfeeding. WOCBP must agree to use a highly effective method of contraception during the study and for 28 days after the last injection of the study drug.
7. Male subjects who are able to father a child must agree to avoid impregnating a partner, to adhere to a highly effective method of contraception and to not donate sperm during the study and for 28 days after the last injection of the study drug.

Exclusion Criteria: Part 1

Patients are excluded from the study if any of the following criteria apply:

1. Unlikely to comply with protocol procedures, restrictions and requirements as judged by the Investigator.
2. Known pregnancy or breastfeeding.
3. Any PET scan done within 10 physical half-lives of the PET agent prior to receiving study intervention.
4. Patients participating in another clinical trial at the time of screening for this study.
5. Patients who have had systemic anti-cancer therapy administered in the 14 days prior to IP administration.
6. Has undergone or plans to undergo PET or single-photon emission computerized tomography (SPECT) imaging with any other FAPi imaging agent within 6 months prior to or after participating in this trial.
7. History of QT/QTc interval prolongation, a marked baseline QT/QTc interval prolongation (e.g., repeated demonstration of a QTc interval, calculated with Fridericia's correction, > 450 milliseconds) or taking medication known to cause QT/QTc prolongation.
8. A history of additional risk factors for Torsades de Pointes (e.g., heart failure, hypokalemia, family history of long QT syndrome).

Exclusion Criteria: Part 2

1. Patients who have had neoadjuvant anti-cancer therapy administered in the 14 days prior to IP administration.
2. Evidence of metastatic or advanced, inoperable disease.
3. Unlikely to comply with protocol procedures, restrictions and requirements and judged by the investigator to be unsuitable for participation.
4. Known pregnancy or breastfeeding.
5. Any PET scan done within 10 physical half-lives of the PET agent prior to receiving study intervention.
6. Patients participating in another clinical trial at the time of screening for this study.
7. Has undergone or plans to undergo PET or SPECT imaging with any other FAPi imaging agent within 6 months prior to or after participating in this trial.
8. History of QT/QTc interval prolongation, a marked baseline QT/QTc interval prolongation (e.g., repeated demonstration of a QTc interval, calculated with Fridericia's correction, > 450 milliseconds) or taking drugs known to cause QT/QTc prolongation.
9. A history of additional risk factors for Torsades de Pointes (e.g., heart failure, hypokalemia, family history of long QT syndrome

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Primary Part 1 Biodistribution of 64Cu-LNTH-1363S | During serial PET/CT scans taken on Day 1 at the following timepoints at 0.5 hour ± 10 minutes, 1 hour ±10 minutes, 2 hours ± 15 minutes, 4 to 6 hours, and 24 hours ± 4 hours post study intervention administration.
  Time Activity Curves (TACs) describing percentage of the injected activity versus time will be derived for selected organs and tumor lesions and absorbed radiation doses of 64Cu-LNTH-1363S in critical organs (e.g., kidneys, liver) will be estimated.
Primary Part 1 - Optimal dose (radioactivity) and imaging time window of 64Cu-LNTH-1363S | During serial PET/CT scans taken on Day 1 at the following timepoints at 0.5 hour ± 10 minutes, 1 hour ±10 minutes, 2 hours ± 15 minutes, 4 to 6 hours, and 24 hours ± 4 hours post study intervention administration.
  Optimal dose (radioactivity) and imaging time window will be determined by using image quality scores from blinded central reviews. Each patient will receive 8 ± 1 mCi of 64Cu-LNTH-1363S. The raw data of each patient PET scan will be re-processed using a computer program to simulate scans of the same patient with lower injected activities (6 mCi and 4 mCi).
Primary Part 2 - Correlation of 64Cu-LNTH-1363S biodistribution with Immunohistochemistry FAP expression | Post surgery tissue collection to end of study
  Correlation of 64Cu-LNTH-1363S biodistribution with FAP expression by IHC (SUVmean and SUVmax vs IHC score) and compare to circulating FAP in blood as analyzed by ELISA method.

SECONDARY OUTCOMES:
Secondary Parts 1 and 2 Safety and Tolerability | Part1: From IP administration until the Day 7 (± 1 day) telephone follow up. Part 2: From time of IP administration to until post-surgery IHC sample collection.
  Safety and tolerability profile of 64Cu-LNTH-1363S in patients with sarcoma and GITs based on:
  * Frequency and severity of adverse events (AEs) and serious AEs (SAEs) measured by Common Terminology Criteria for AEs (CTCAE) v5.0 or higher.
  * Changes in vital signs
  * Changes in laboratory parameters
  * Changes in electrocardiogram (ECG)parameters
    • Exposure-response relationships:
  * Relationship of AEs to exposure (dose and concentrations).
Secondary Part 1 FAP expression profile of 64Cu-LNTH-1363S in patients with sarcoma | From Day 1 until the end of the Scheduled Surgery: IHC sample collection
  Correlation of 64Cu-LNTH-1363S biodistribution with FAP expression by immunohistochemistry (IHC) (SUVmean and SUVmax vs IHC score) and compare to circulating FAP in blood as analyzed by ELISA method.
Secondary Part 1 and Part 2 Cardiac Safety | Continuous ECG monitoring at Visit 2
  Monitor cardiac safety and look for signals suggesting a concentration-response relationship of 64Cu-LNTH-1363S for QT/corrected QT interval (QTc) prolongation.
Secondary Part 2 Validate optimal radioactivity in patients with sarcoma or GIT cancer | From start of Part 2 to 6 patients enrolled with qualifying imaging
  Validate optimal radioactivity in patients with sarcoma or GIT cancer, if the optimal radioactivity determined in Part 1 is less than 8 ± 1 mCi. Validation to be completed on image quality score of first 6 patients, if optimal radioactivity determined in Part 1 is less than 8 ± 1 mCi.

OTHER OUTCOMES:
Exploratory Part 1 and Part 2 | From post study intervention administration imaging in each patient (0.5 hour ± 10 minutes, 1 hour ±10 minutes, 2 hours ± 15 minutes, 4 to 6 hours, and 24 hours ± 4 hours in Part 1 and 2 timepoints in Part 2) to the end of the study].
  Develop an AI system for detecting and characterizing cancer lesion(s) expressing FAP using 64Cu-LNTH-1363S, through Correlation between automated measurement of physiological uptake of 64Cu-LNTH-1363S with manual measurement results; and through the determination of the detection rate of possible site of cancer lesion(s) with 64Cu-LNTH-1363S using an AI enabled reading system when compared to central reader assessments.
  Part 2: Estimation of total tumor burden using an AI enabled reading system.
Correlation between LRRC15 IHC and FAP expression | Availability of tumor tissue will be assessed at Screening visit.
  Correlation of LRRC15 expression to 64Cu-LNTH-1363S biodistribution and FAP expression (determined by IHC)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - City of Hope, Duarte, California
  - UC Irvine Health - Chao Family Comprehensive Cancer Center, Orange, California
  - Stanford Hospital & Clinics, Stanford, California
  - BAMF Health, Inc., Grand Rapids, Michigan
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio